CLINICAL TRIAL: NCT03483961
Title: A Phase 2 Parallel-Group, Randomized, Double-Blind Study to Assess the Safety and Immunogenicity of PXVX0317 (Chikungunya Virus Virus-Like Particle Vaccine [CHIKV-VLP], Unadjuvanted or Alum-adjuvanted)
Brief Title: Trial of a Chikungunya Vaccine, PXVX0317 CHIKV-VLP, in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PXVX-CV-317-001
Record Dates: First submitted 2018-03-16; First posted 2018-03-30 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Group 1: 20 mcg/unadjuvanted (Day 1 & 29) (Experimental): 20 mcg CHIKV VLP/unadjuvanted (Day 1) // Placebo (Day 15) // 20 mcg CHIKV VLP/unadjuvanted (Day 29)
  Interventions: Biological: CHIKV VLP/unadjuvanted; Biological: Placebo
- Group 2: 6 mcg/adjuvanted (Day 1 & 29) (Experimental): 6 mcg CHIKV VLP/adjuvanted (Day 1) // Placebo (Day 15) // 6 mcg CHIKV VLP/adjuvanted (Day 29)
  Interventions: Biological: CHIKV VLP/adjuvanted; Biological: Placebo
- Group 3: 10 mcg/adjuvanted (Day 1 & 29) (Experimental): 10 mcg CHIKV VLP/adjuvanted (Day 1) // Placebo (Day 15) // 10 mcg CHIKV VLP/adjuvanted (Day 29)
  Interventions: Biological: CHIKV VLP/adjuvanted; Biological: Placebo
- Group 4: 20mcg/adjuvanted (Day 1 & 29);40mcg/adjuvant (Day 547) (Experimental): 20 mcg CHIKV VLP/adjuvanted (Day 1) // Placebo (Day 15) // 20 mcg CHIKV VLP/adjuvanted (Day 29) // 40 mcg CHIKV (Day 547)
  Interventions: Biological: CHIKV VLP/adjuvanted; Biological: Placebo
- Group 5: 6 mcg/adjuvanted (Day 15 & 29) (Experimental): Placebo (Day 1) // 6 mcg CHIKV VLP/adjuvanted (Day 15) // 6 mcg CHIKV VLP/adjuvanted (Day 29)
  Interventions: Biological: CHIKV VLP/adjuvanted; Biological: Placebo
- Group 6: 10 mcg/adjuvanted (Day 15 & 29) (Experimental): Placebo (Day 1) // 10 mcg CHIKV VLP/adjuvanted (Day 15) // 10 mcg CHIKV VLP/adjuvanted (Day 29)
  Interventions: Biological: CHIKV VLP/adjuvanted; Biological: Placebo
- Group 7: 20 mcg/adjuvanted (Day 15 & 29) (Experimental): Placebo (Day 1) // 20 mcg CHIKV VLP/adjuvanted (Day 15) // 20 mcg CHIKV VLP/adjuvanted (Day 29)
  Interventions: Biological: CHIKV VLP/adjuvanted; Biological: Placebo
- Group 8: 40 mcg/adjuvanted (Day 29) (Experimental): Placebo (Day 1) // Placebo (Day 15) // 40 mcg CHIKV VLP/adjuvanted (Day 29)
  Interventions: Biological: CHIKV VLP/adjuvanted; Biological: Placebo
- Group 9: 20 mcg/adjuvanted (Day 1 & 29) (Experimental): 20 mcg CHIKV VLP/adjuvanted (Day 1) // 20 mcg CHIKV VLP/adjuvanted (Day 29). This group will also have plasmapheresis performed on Day 57 and Leukapheresis on Day 182
  Interventions: Biological: CHIKV VLP/adjuvanted
- Group 10: 40 mcg/adjuvanted (Day 1) (Experimental): 40 mcg CHIKV VLP/adjuvanted (Day 1). This group will also have plasmapheresis performed on Day 22.
  Interventions: Biological: CHIKV VLP/adjuvanted

INTERVENTIONS:
Biological: CHIKV VLP/unadjuvanted — Vaccine consists of virus-like particles of chikungunya virus antigens
  Arms: Group 1: 20 mcg/unadjuvanted (Day 1 & 29)
Biological: CHIKV VLP/adjuvanted — Adjuvanted formulation includes Alhydrogel
  Arms: Group 10: 40 mcg/adjuvanted (Day 1); Group 2: 6 mcg/adjuvanted (Day 1 & 29); Group 3: 10 mcg/adjuvanted (Day 1 & 29); Group 4: 20mcg/adjuvanted (Day 1 & 29);40mcg/adjuvant (Day 547); Group 5: 6 mcg/adjuvanted (Day 15 & 29); Group 6: 10 mcg/adjuvanted (Day 15 & 29); Group 7: 20 mcg/adjuvanted (Day 15 & 29); Group 8: 40 mcg/adjuvanted (Day 29); Group 9: 20 mcg/adjuvanted (Day 1 & 29)
Biological: Placebo — Placebo is vaccine diluent alone
  Arms: Group 1: 20 mcg/unadjuvanted (Day 1 & 29); Group 2: 6 mcg/adjuvanted (Day 1 & 29); Group 3: 10 mcg/adjuvanted (Day 1 & 29); Group 4: 20mcg/adjuvanted (Day 1 & 29);40mcg/adjuvant (Day 547); Group 5: 6 mcg/adjuvanted (Day 15 & 29); Group 6: 10 mcg/adjuvanted (Day 15 & 29); Group 7: 20 mcg/adjuvanted (Day 15 & 29); Group 8: 40 mcg/adjuvanted (Day 29)

SUMMARY:
The goal of this Phase 2 trial is to evaluate the immune response to and safety profile of various doses/formulations/and schedules of administration of PXVX0317 in healthy adults.

Primary Objective:

To assess the immune response to the vaccine

Secondary Objectives:

To assess the kinetics of the immune response to different doses/formulations/schedules To assess the persistence of immune responses to different doses/formulations/schedules To assess the effect of a booster dose of the vaccine

Safety Objective:

To assess local and systemic reactions to the vaccine and to describe the safety profile of the vaccine

DETAILED DESCRIPTION:
The trial will explore 8 formulation/schedule combinations of CHIKV VLP vaccine with or without Alhydrogel adjuvant, and will also explore different dose schedules of Day 1 and 15 or Day 1 and 29 or Day 29 only.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18 to 45 years old (inclusive)
3. Using an acceptable method of contraception (if female of childbearing potential).
4. Able and willing to provide informed consent for study participation.

Exclusion Criteria:

1. Current acute febrile illness.
2. Clinically significant cardiac, respiratory, or rheumatologic disease, in the opinion of the Investigator.
3. Pregnant or breast-feeding.
4. Laboratory evidence of infection with Hepatitis B/C or HIV.
5. History of chikungunya virus infection.
6. Travel to a World Health Organization-designated chikungunya-endemic region within 30 days prior to Day 1.
7. History of allergic reaction to any component of CHIKV-VLP vaccine, Diluent, or Alhydrogel®.
8. Inability to discontinue systemic immunomodulatory or immunosuppressive medications 30 days prior to Day 1.
9. Received or plans to receive any licensed vaccine from 30 days prior to Day 1 through Day 57.
10. Received or plans to receive an investigational agent from 30 days prior to Day 1 through the duration of study participation.
11. Any other condition that, in the opinion of the Investigator, creates an unacceptable risk to the subject.
12. Any other condition that, in the opinion of the Investigator, may interfere with the conduct of the study or the validity of the data.
13. Any other condition that, in the opinion of the Investigator, creates an unacceptable safety risk for apheresis (Group 9 & 10 only).
14. Restricted venous access that would prevent the collection of PBMCs, plasma, and lymphocytes necessary for participation (Group 9 & 10 only).
15. Weight < 110 pounds (Group 9 & 10 only)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 445 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarty, MD, Study Director — Emergent BioSolutions
Locations (3):
- United States (3):
  - Johnson County Clin-Trials, Lenexa, Kansas
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennett SR, McCarty JM, Ramanathan R, Mendy J, Richardson JS, Smith J, Alexander J, Ledgerwood JE, de Lame PA, Royalty Tredo S, Warfield KL, Bedell L. Safety and immunogenicity of PXVX0317, an aluminium hydroxide-adjuvanted chikungunya virus-like particle vaccine: a randomised, double-blind, parallel-group, phase 2 trial. Lancet Infect Dis. 2022 Sep;22(9):1343-1355. doi: 10.1016/S1473-3099(22)00226-2. Epub 2022 Jun 13. PMID 35709798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 3 U.S. sites.
Groups:
- Group 1: 20 mcg/Unadjuvant (Day 1 & 29): 20 mcg CHIKV VLP/unadjuvanted (Day 1) // Placebo (Day 15) // 20 mcg CHIKV VLP/unadjuvanted (Day 29)
  CHIKV VLP/unadjuvanted: Vaccine consists of virus-like particles of chikungunya virus antigens
  Placebo: Placebo is vaccine diluent alone
- Group 2: 6 mcg/Adjuvant (Day 1 & 29): 6 mcg CHIKV VLP/adjuvanted (Day 1) // Placebo (Day 15) // 6 mcg CHIKV VLP/adjuvanted (Day 29)
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
  Placebo: Placebo is vaccine diluent alone
- Group 3: 10 mcg/Adjuvant (Day 1 & 29): 10 mcg CHIKV VLP/adjuvanted (Day 1) // Placebo (Day 15) // 10 mcg CHIKV VLP/adjuvanted (Day 29)
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
  Placebo: Placebo is vaccine diluent alone
- Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547): 20 mcg CHIKV VLP/adjuvanted (Day 1) // Placebo (Day 15) // 20 mcg CHIKV VLP/adjuvanted (Day 29) // 40 mcg CHIKV (Day 547)
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
  Placebo: Placebo is vaccine diluent alone
- Group 5: 6 mcg/Adjuvant (Day 15 & 29): Placebo (Day 1) // 6 mcg CHIKV VLP/adjuvanted (Day 15) // 6 mcg CHIKV VLP/adjuvanted (Day 29)
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
  Placebo: Placebo is vaccine diluent alone
- Group 6: 10 mcg/Adjuvant (Day 15 & 29): Placebo (Day 1) // 10 mcg CHIKV VLP/adjuvanted (Day 15) // 10 mcg CHIKV VLP/adjuvanted (Day 29)
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
  Placebo: Placebo is vaccine diluent alone
- Group 7: 20 mcg/Adjuvant (Day 15 & 29): Placebo (Day 1) // 20 mcg CHIKV VLP/adjuvanted (Day 15) // 20 mcg CHIKV VLP/adjuvanted (Day 29)
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
  Placebo: Placebo is vaccine diluent alone
- Group 8: 40 mcg/Adjuvant (Day 29): Placebo (Day 1) // Placebo (Day 15) // 40 mcg CHIKV VLP/adjuvanted (Day 29)
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
  Placebo: Placebo is vaccine diluent alone
- Group 9: 20 mcg/Adjuvant (Day 1 & 29): 20 mcg CHIKV VLP/adjuvanted (Day 1) // 20 mcg CHIKV VLP/adjuvanted (Day 29). This group will also have plasmapheresis performed on Day 57 and Leukapheresis on Day 182
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
- Group 10: 40 mcg/Adjuvant (Day 1): 40 mcg CHIKV VLP/adjuvanted (Day 1). This group will also have plasmapheresis performed on Day 22.
  CHIKV VLP/adjuvanted: Adjuvanted formulation includes Alhydrogel
Period: Overall Study
Arm/Group | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) | Group 8: 40 mcg/Adjuvant (Day 29) | Group 9: 20 mcg/Adjuvant (Day 1 & 29) | Group 10: 40 mcg/Adjuvant (Day 1)
Started | 53 | 52 | 51 | 50 | 53 | 53 | 51 | 52 | 20 | 10
Exposed / Safety | 53 | 52 | 50 (One subject was randomized to Group 3 but treated in Group 4 due to a dispensing error.) | 51 (One subject was randomized to Group 3 but treated in Group 4 due to a dispensing error.) | 53 (One subject did not receive PXVX0317 but is in the Exposed / Safety population because of receipt of placebo.) | 53 | 51 (One subject did not receive PXVX0317 but is in the Exposed / Safety population because of receipt of placebo.) | 52 (Two subjects did not receive PXVX0317 but are in the Exposed / Safety population because of receipt of placebo.) | 20 | 10
Immunogenicity-evaluable | 47 | 44 | 44 | 45 | 48 | 48 | 47 | 50 | 20 | 10
Completed | 42 | 42 | 39 | 41 | 43 | 47 | 46 | 39 | 18 | 10
Not Completed | 11 | 10 | 12 | 9 | 10 | 6 | 5 | 13 | 2 | 0
Not completed — Lost to Follow-up | 7 | 6 | 6 | 6 | 6 | 4 | 4 | 11 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 5 | 3 | 4 | 2 | 1 | 2 | 1 | 0
Not completed — Other than AE, death, PI decision, LTFU, noncompliance, study terminated, or withdrawal of consent | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) | Group 8: 40 mcg/Adjuvant (Day 29) | Group 9: 20 mcg/Adjuvant (Day 1 & 29) | Group 10: 40 mcg/Adjuvant (Day 1) | Total
Number analyzed (Participants) | 53 | 52 | 51 | 50 | 53 | 53 | 51 | 52 | 20 | 10 | 445
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5
  Between 18 and 65 years | 50 | 51 | 51 | 50 | 53 | 52 | 51 | 52 | 20 | 10 | 440
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (8.22) | 31.2 (8.26) | 31.2 (7.64) | 33.7 (7.53) | 30.6 (7.72) | 32.9 (7.53) | 32.4 (7.78) | 31.6 (7.82) | 27.1 (7.58) | 29.6 (7.65) | 31.5 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 37 | 32 | 38 | 29 | 27 | 26 | 7 | 3 | 259
  Male | 23 | 22 | 14 | 18 | 15 | 24 | 24 | 26 | 13 | 7 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 4 | 3 | 4 | 8 | 2 | 4 | 2 | 1 | 35
  Not Hispanic or Latino | 50 | 48 | 47 | 47 | 49 | 45 | 49 | 48 | 18 | 9 | 410
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Asian | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Black or African American | 10 | 9 | 14 | 13 | 14 | 9 | 15 | 7 | 7 | 6 | 104
  White | 43 | 40 | 36 | 35 | 36 | 40 | 34 | 41 | 11 | 4 | 320
  More than one race | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 52 | 51 | 50 | 53 | 53 | 51 | 52 | 20 | 10 | 445
Day 1 predose (baseline) geometric mean anti-chikungunya luciferase neutralizing antibody titer. [Geometric Mean (Full Range); unit: titer] — Day 1 predose (baseline) geometric mean anti-chikungunya luciferase neutralizing antibody titer. Values below the lower limit of quantitation of 15 were imputed as half the lower limit of quantitation or 7.5. Population: Immunogenicity-evaluable: Exposed participants as treated per protocol (no major protocol deviation or exclusion reason prior to unblinding, all doses received, no prohibited medication, and evaluable serum samples within required time frames).
  titer
    number analyzed (Participants) | 47 | 44 | 44 | 45 | 48 | 48 | 47 | 50 | 20 | 10 | 403
    (all) | 7.5 [7.5 to 7.5] | 7.5 [7.5 to 7.5] | 7.5 [7.5 to 7.5] | 7.5 [7.5 to 7.5] | 7.8 [7.5 to 50.3] | 7.5 [7.5 to 7.5] | 7.5 [7.5 to 7.5] | 7.5 [7.5 to 7.5] | 8.6 [7.5 to 117.1] | 9.0 [7.5 to 46.1] | 7.6 [7.5 to 117.1]

OUTCOME MEASURES:

1. Primary Outcome: Anti-CHIKV Neutralizing Antibody Geometric Mean Titer 28 Days After the Last Injection for Groups 2-8.
Description: To assess the induction of anti-chikungunya virus (CHIKV) neutralizing antibody geometric mean titers by different formulations and schedules, as measured at 28 days after the last injection (Day 57) for Groups 2-8.
Time Frame: Day 57 (from Day 1 vaccination), 28 days after the last injection.
Population: Immunogenicity-evaluable: Exposed participants as treated per protocol (no major protocol deviation or exclusion reason prior to unblinding, all doses received, no prohibited medication, and evaluable serum samples within required time frames).
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) | Group 8: 40 mcg/Adjuvant (Day 29)
Number analyzed (Participants) | 47 | 44 | 44 | 45 | 48 | 48 | 47 | 50
titer | 2057.0 [1584.8 to 2670.0] | 1116.2 [852.5 to 1461.4] | 1465.3 [1119.1 to 1918.4] | 2023.8 [1550.5 to 2641.7] | 920.1 [710.9 to 1190.9] | 1206.9 [932.4 to 1562.2] | 1562.8 [1204.1 to 2028.3] | 1712.5 [1330.0 to 2205.0]
Statistical Analysis 1: Comparison: Group 1: 20 mcg/Unadjuvant (Day 1 & 29) vs Group 2: 6 mcg/Adjuvant (Day 1 & 29) vs Group 3: 10 mcg/Adjuvant (Day 1 & 29) vs Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) vs Group 5: 6 mcg/Adjuvant (Day 15 & 29) vs Group 6: 10 mcg/Adjuvant (Day 15 & 29) vs Group 7: 20 mcg/Adjuvant (Day 15 & 29) vs Group 8: 40 mcg/Adjuvant (Day 29); Groups 2-8 are compared to Group 1; Test type: Superiority; p = 0.0015, ANOVA — All tests were carried out at a 2-sided significance level of 0.05 and no adjustment for multiplicity was applied, since the goal was to rank different formulations rather than to establish inferential values; ANOVA model including site and treatment group as fixed effects assuming normality of log titers. P-value is for Group 2 vs. Group 1
Statistical Analysis 2: Comparison: Group 1: 20 mcg/Unadjuvant (Day 1 & 29) vs Group 2: 6 mcg/Adjuvant (Day 1 & 29) vs Group 3: 10 mcg/Adjuvant (Day 1 & 29) vs Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) vs Group 5: 6 mcg/Adjuvant (Day 15 & 29) vs Group 6: 10 mcg/Adjuvant (Day 15 & 29) vs Group 7: 20 mcg/Adjuvant (Day 15 & 29) vs Group 8: 40 mcg/Adjuvant (Day 29); Groups 2-8 are compared to Group 1; Test type: Superiority; p = 0.0761, ANOVA — [p-value comment as in outcome 1, analysis 1]; ANOVA model including site and treatment group as fixed effects assuming normality of log titers. P-value is for Group 3 vs. Group 1
Statistical Analysis 3: Comparison: Group 1: 20 mcg/Unadjuvant (Day 1 & 29) vs Group 2: 6 mcg/Adjuvant (Day 1 & 29) vs Group 3: 10 mcg/Adjuvant (Day 1 & 29) vs Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) vs Group 5: 6 mcg/Adjuvant (Day 15 & 29) vs Group 6: 10 mcg/Adjuvant (Day 15 & 29) vs Group 7: 20 mcg/Adjuvant (Day 15 & 29) vs Group 8: 40 mcg/Adjuvant (Day 29); Groups 2-8 are compared to Group 1; Test type: Superiority; p = 0.9317, ANOVA — [p-value comment as in outcome 1, analysis 1]; ANOVA model including site and treatment group as fixed effects assuming normality of log titers. P-value is for Group 4 vs. Group 1
Statistical Analysis 4: Comparison: Group 1: 20 mcg/Unadjuvant (Day 1 & 29) vs Group 2: 6 mcg/Adjuvant (Day 1 & 29) vs Group 3: 10 mcg/Adjuvant (Day 1 & 29) vs Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) vs Group 5: 6 mcg/Adjuvant (Day 15 & 29) vs Group 6: 10 mcg/Adjuvant (Day 15 & 29) vs Group 7: 20 mcg/Adjuvant (Day 15 & 29) vs Group 8: 40 mcg/Adjuvant (Day 29); Groups 2-8 are compared to Group 1; Test type: Superiority; p < .0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; ANOVA model including site and treatment group as fixed effects assuming normality of log titers. P-value is for Group 5 vs. Group 1
Statistical Analysis 5: Comparison: Group 1: 20 mcg/Unadjuvant (Day 1 & 29) vs Group 2: 6 mcg/Adjuvant (Day 1 & 29) vs Group 3: 10 mcg/Adjuvant (Day 1 & 29) vs Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) vs Group 5: 6 mcg/Adjuvant (Day 15 & 29) vs Group 6: 10 mcg/Adjuvant (Day 15 & 29) vs Group 7: 20 mcg/Adjuvant (Day 15 & 29) vs Group 8: 40 mcg/Adjuvant (Day 29); Groups 2-8 are compared to Group 1; Test type: Superiority; p = 0.0045, ANOVA — [p-value comment as in outcome 1, analysis 1]; ANOVA model including site and treatment group as fixed effects assuming normality of log titers. P-value is for Group 6 vs. Group 1
Statistical Analysis 6: Comparison: Group 1: 20 mcg/Unadjuvant (Day 1 & 29) vs Group 2: 6 mcg/Adjuvant (Day 1 & 29) vs Group 3: 10 mcg/Adjuvant (Day 1 & 29) vs Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) vs Group 5: 6 mcg/Adjuvant (Day 15 & 29) vs Group 6: 10 mcg/Adjuvant (Day 15 & 29) vs Group 7: 20 mcg/Adjuvant (Day 15 & 29) vs Group 8: 40 mcg/Adjuvant (Day 29); Groups 2-8 are compared to Group 1; Test type: Superiority; p = 0.1437, ANOVA — [p-value comment as in outcome 1, analysis 1]; ANOVA model including site and treatment group as fixed effects assuming normality of log titers. P-value is for Group 7 vs. Group 1
Statistical Analysis 7: Comparison: Group 1: 20 mcg/Unadjuvant (Day 1 & 29) vs Group 2: 6 mcg/Adjuvant (Day 1 & 29) vs Group 3: 10 mcg/Adjuvant (Day 1 & 29) vs Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) vs Group 5: 6 mcg/Adjuvant (Day 15 & 29) vs Group 6: 10 mcg/Adjuvant (Day 15 & 29) vs Group 7: 20 mcg/Adjuvant (Day 15 & 29) vs Group 8: 40 mcg/Adjuvant (Day 29); Groups 2-8 are compared to Group 1; Test type: Superiority; p = 0.3216, ANOVA — [p-value comment as in outcome 1, analysis 1]; ANOVA model including site and treatment group as fixed effects assuming normality of log titers. P-value is for Group 8 vs. Group 1

2. Secondary Outcome: Kinetics of Anti-chikungunya Virus (CHIKV) Neutralizing Antibody Geometric Mean Titer for Groups 2-8.
Description: To describe the kinetics of induction of anti-CHIKV neutralizing antibody geometric mean titers by different formulations and schedules for Groups 2-8.
Time Frame: At Days 8, 15, 22, 29, 36, and 57.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) | Group 8: 40 mcg/Adjuvant (Day 29)
Number analyzed (Participants) | 47 | 44 | 44 | 45 | 48 | 48 | 47 | 50
titer
  Day 8: number analyzed (Participants) | 47 | 43 | 44 | 44 | 47 | 47 | 47 | 49
  Day 8 | 70.6 [53.2 to 93.7] | 34.3 [25.6 to 46.1] | 72.6 [54.2 to 97.2] | 117.6 [87.8 to 157.4] | 8.4 [6.3 to 11.1] | 7.5 [5.7 to 10.0] | 7.5 [5.7 to 10.0] | 7.5 [5.7 to 9.9]
  Day 15 | 419.3 [323.6 to 543.4] | 189.4 [144.9 to 247.6] | 530.2 [405.6 to 693.0] | 912.7 [700.4 to 1189.5] | 7.7 [6.0 to 10.0] | 7.5 [5.8 to 9.7] | 7.7 [5.9 to 9.9] | 7.5 [5.8 to 9.6]
  Day 22 | 691.5 [499.2 to 957.9] | 351.3 [250.9 to 492.0] | 1400.2 [999.9 to 1960.8] | 2198.1 [1575.6 to 3066.5] | 46.4 [33.6 to 64.1] | 63.1 [45.7 to 87.1] | 119.0 [85.9 to 164.9] | 7.5 [5.5 to 10.3]
  Day 29 | 417.2 [305.4 to 570.0] | 277.3 [200.9 to 382.8] | 890.5 [645.1 to 1229.2] | 1238.1 [900.2 to 1702.9] | 258.0 [189.5 to 351.3] | 328.8 [241.5 to 447.6] | 886.2 [648.7 to 1210.5] | 8.2 [6.0 to 11.0]
  Day 36: number analyzed (Participants) | 47 | 44 | 44 | 45 | 48 | 48 | 46 | 50
  Day 36 | 3442.8 [2533.9 to 4677.8] | 1675.8 [1220.9 to 2300.2] | 2772.4 [2019.8 to 3805.4] | 3435.0 [2511.4 to 4698.1] | 1327.7 [980.4 to 1797.9] | 2155.4 [1591.6 to 2919.0] | 3609.0 [2647.7 to 4919.3] | 157.9 [117.3 to 212.6]
  Day 57 | 2057.0 [1584.8 to 2670.0] | 1116.2 [852.5 to 1461.4] | 1465.3 [1119.1 to 1918.4] | 2023.8 [1550.5 to 2641.7] | 920.1 [710.9 to 1190.9] | 1206.9 [932.4 to 1562.2] | 1562.8 [1204.1 to 2028.3] | 1712.5 [1330.0 to 2205.0]

3. Secondary Outcome: Differences in Persistence of Neutralizing Antibody Geometric Mean Titer for Groups 2-8.
Description: To assess differences in persistence of neutralizing antibody geometric mean titers induced by different formulations and schedules, as measured up to 731 days after the last injection (Day 760) relative to earlier time points for Groups 2-8.
Time Frame: At Days 182, 365, 547, and 760.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) | Group 8: 40 mcg/Adjuvant (Day 29)
Number analyzed (Participants) | 47 | 44 | 44 | 45 | 48 | 48 | 47 | 50
titer
  Day 182: number analyzed (Participants) | 46 | 40 | 39 | 43 | 44 | 46 | 47 | 48
  Day 182 | 345.1 [258.1 to 461.3] | 209.0 [153.1 to 285.2] | 358.4 [261.6 to 491.2] | 486.6 [360.5 to 656.9] | 253.4 [188.4 to 340.9] | 303 [226.7 to 405.0] | 388.1 [291.3 to 517.1] | 505.7 [380.7 to 671.8]
  Day 365: number analyzed (Participants) | 42 | 38 | 36 | 42 | 41 | 43 | 43 | 46
  Day 365 | 243.4 [176.8 to 334.9] | 137.5 [98.3 to 192.3] | 226.7 [160.6 to 320.0] | 336.6 [244.6 to 463.2] | 195.2 [141.3 to 269.6] | 246.9 [180.1 to 338.4] | 302.0 [220.3 to 414.0] | 491.7 [362.5 to 667.0]
  Day 547: number analyzed (Participants) | 41 | 44 | 44 | 41 | 48 | 48 | 47 | 40
  Day 547 | 169.2 [126.2 to 226.8] | NA [NA to NA] — Follow-up to Day 365 in this group. | NA [NA to NA] — Follow-up to Day 365 in this group. | 215.7 [160.9 to 289.1] | NA [NA to NA] — Follow-up to Day 365 in this group. | NA [NA to NA] — Follow-up to Day 365 in this group. | NA [NA to NA] — Follow-up to Day 365 in this group. | 297.9 [221.4 to 400.8]
  Day 760: number analyzed (Participants) | 40 | 44 | 44 | 39 | 48 | 48 | 47 | 38
  Day 760 | 169.8 [122.4 to 235.5] | NA [NA to NA] — Follow-up to Day 365 in this group. | NA [NA to NA] — Follow-up to Day 365 in this group. | 5365.1 [3853.2 to 7470.1] | NA [NA to NA] — Follow-up to Day 365 in this group. | NA [NA to NA] — Follow-up to Day 365 in this group. | NA [NA to NA] — Follow-up to Day 365 in this group. | 279.7 [200.1 to 391.1]

4. Secondary Outcome: Boosting of Vaccine-induced Neutralizing Antibody Geometric Mean Titer by a Booster Dose of PXVX0317 for Group 4 Only.
Description: To assess the effect of a booster dose of PXVX0317 on neutralizing antibody geometric mean titers when given at Day 547 for Group 4 only. Antibody levels will be measured at Day 547 prior to the booster dose and again 28 days later on Day 575 and then at Day 760.
Time Frame: Antibody levels will be measured at Day 547 prior to the booster dose and again 28 days later on Day 575 and then at Day 760.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547)
Number analyzed (Participants) | 47
titer
  Day 547 (pre-boost): number analyzed (Participants) | 39
  Day 547 (pre-boost) | 223.6 [166.7 to 299.9]
  Day 575 (post-boost): number analyzed (Participants) | 38
  Day 575 (post-boost) | 12325.8 [8951.4 to 16972.4]
  Day 760 (post-boost): number analyzed (Participants) | 38
  Day 760 (post-boost) | 5874.2 [4269.4 to 8082.3]

5. Secondary Outcome: Percentage of Participants With an Anti-CHIKV Neutralizing Antibody Titer Exceeding the Following Cutoff Values: ≥15, 40, 160, 640, and 4-fold Rise Over Baseline.
Description: Percentage of participants with an anti-CHIKV neutralizing antibody titer exceeding the following cutoff values: ≥15, 40, 160, 640, and 4-fold rise over baseline.
Time Frame: Day 57 (from Day 1 vaccination), 28 days after the last injection.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) | Group 8: 40 mcg/Adjuvant (Day 29)
Number analyzed (Participants) | 47 | 44 | 44 | 45 | 48 | 48 | 47 | 50
Participants
  Titer at or above 15 | 47 | 44 | 44 | 45 | 48 | 48 | 47 | 50
  Titer at or above 40 | 47 | 44 | 43 | 45 | 48 | 48 | 47 | 50
  Titer at or above 160 | 47 | 42 | 43 | 45 | 47 | 48 | 46 | 50
  Titer at or above 640 | 43 | 32 | 41 | 43 | 29 | 40 | 41 | 44
  Titer at or above 4-fold rise over baseline | 47 | 44 | 43 | 45 | 48 | 48 | 47 | 50

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events were monitored through Day 760 (Groups 1, 4, and 8), Day 365 (Groups 2, 3, 5, 6, and 7), Day 182 (Group 9), and Day 29 (Group 10), but only unsolicited adverse events occurring through Day 57 (end of treatment and observation period, 28 days after last dose for Groups 1-8) are reported.
Description: One subject was randomized to Group 3 but treated in Group 4 due to a dispensing error. This participant was counted in Group 3 in the Participant Flow Number Started but was counted in Group 4 for the safety population for all safety analyses.
Arm/Group | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) | Group 8: 40 mcg/Adjuvant (Day 29) | Group 9: 20 mcg/Adjuvant (Day 1 & 29) | Group 10: 40 mcg/Adjuvant (Day 1)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52 | 0/50 | 0/51 | 0/53 | 0/53 | 0/51 | 0/52 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/52 | 2/50 | 1/51 | 0/53 | 0/53 | 2/51 | 3/52 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 26/53 | 35/52 | 36/50 | 34/51 | 29/53 | 28/53 | 30/51 | 34/52 | 12/20 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) (N=53) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) (N=52) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) (N=50) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) (N=51) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) (N=53) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) (N=53) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) (N=51) | Group 8: 40 mcg/Adjuvant (Day 29) (N=52) | Group 9: 20 mcg/Adjuvant (Day 1 & 29) (N=20) | Group 10: 40 mcg/Adjuvant (Day 1) (N=10)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Induced abortion haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 20 mcg/Unadjuvant (Day 1 & 29) (N=53) | Group 2: 6 mcg/Adjuvant (Day 1 & 29) (N=52) | Group 3: 10 mcg/Adjuvant (Day 1 & 29) (N=50) | Group 4: 20mcg/Adjuvant(Day 1 & 29);40mcg/Adjuvant (Day 547) (N=51) | Group 5: 6 mcg/Adjuvant (Day 15 & 29) (N=53) | Group 6: 10 mcg/Adjuvant (Day 15 & 29) (N=53) | Group 7: 20 mcg/Adjuvant (Day 15 & 29) (N=51) | Group 8: 40 mcg/Adjuvant (Day 29) (N=52) | Group 9: 20 mcg/Adjuvant (Day 1 & 29) (N=20) | Group 10: 40 mcg/Adjuvant (Day 1) (N=10)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 4 (4) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea, solicited (Gastrointestinal disorders) | 8 (9) | 6 (10) | 8 (8) | 14 (17) | 4 (4) | 5 (7) | 6 (6) | 6 (8) | 1 (1) | 0 (0)
Injection site pain, solicited (General disorders) | 19 (25) | 27 (41) | 23 (35) | 29 (63) | 18 (25) | 18 (27) | 18 (30) | 26 (32) | 10 (16) | 2 (2)
Fatigue, solicited (General disorders) | 11 (16) | 12 (18) | 12 (14) | 19 (27) | 7 (7) | 7 (10) | 11 (17) | 10 (15) | 2 (2) | 2 (2)
Malaise, solicited (General disorders) | 7 (8) | 7 (10) | 6 (7) | 14 (15) | 4 (4) | 7 (10) | 10 (13) | 9 (11) | 2 (2) | 1 (1)
Chills, solicited (General disorders) | 1 (1) | 3 (3) | 5 (5) | 8 (9) | 3 (3) | 4 (6) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Myalgia, solicited (Musculoskeletal and connective tissue disorders) | 11 (12) | 12 (15) | 12 (18) | 21 (35) | 11 (14) | 10 (18) | 11 (19) | 11 (11) | 0 (0) | 2 (2)
Arthralgia, solicited (Musculoskeletal and connective tissue disorders) | 3 (4) | 9 (11) | 4 (6) | 12 (16) | 3 (4) | 4 (7) | 4 (8) | 6 (6) | 1 (1) | 1 (1)
Headache, solicited (Nervous system disorders) | 11 (14) | 14 (23) | 18 (21) | 20 (31) | 11 (12) | 11 (17) | 14 (19) | 19 (26) | 3 (4) | 1 (1)
Pyrexia, solicited (General disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or release study data after the earlier of (a) the date of publication of a multi-center publication coordinated by Sponsor on the study data, or (b) the date of submission of the study data by Sponsor to regulatory authorities for regulatory approval; provided that PI furnishes Sponsor with a copy of any proposed publication or release at least ninety days in advance of the proposed submission or presentation date for review. PI must acknowledge Sponsor on any publication.

DOCUMENTS (6):
  • Study Protocol: Protocol Cover Page (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT03483961/Prot_000.pdf
  • Study Protocol: Protocol Cover Page (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT03483961/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Cover Page (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT03483961/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Cover Page (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT03483961/SAP_003.pdf
  • Informed Consent Form: Informed Consent Form Cover page (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03483961/ICF_004.pdf
  • Informed Consent Form: Informed Consent Form Cover page (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03483961/ICF_005.pdf